CLINICAL TRIAL: NCT01037712
Title: In UTERO Treatment of Cytomegalovirus Congenital Infection With Valacyclovir: Prospective Multicenter Randomized Trial Versus Placebo
Brief Title: In UTERO Treatment of Cytomegalovirus Congenital Infection With Valacyclovir
Acronym: CYMEVAL
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: not enough inclusion
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P070115
Record Dates: First submitted 2009-12-21; First posted 2009-12-23 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2011-02

CONDITIONS: Viral Disease; Cytomegalovirus Infection
Keywords: Foetuses infection with CMV; neurological handicap of infectious origin.
MeSH Terms: conditions — Virus Diseases; Cytomegalovirus Infections | interventions — Valacyclovir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ZELITREX (Experimental): ZELITREX
  Interventions: Drug: Valacyclovir (ZELITREX)
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Valacyclovir (ZELITREX) — 2g, 8g/day, 4 a day 23 weeks maximum.
  Arms: ZELITREX
Drug: Placebo — placebo
  Arms: Placebo

SUMMARY:
The infection with cytomegalovirus (CMV) is the first cause of congenital neurological handicap of infectious origin. It is probable that the neonatal viral load is correlated with becoming of infected new-born babies. Among the active antiviral treatments against CMV, valacyclovir is the only whose fetal and maternal tolerance was evaluated during the pregnancy. Its harmlessness and its aptitude to decrease the CMV viral load justify to evaluate it in a study against placebo. Decrease the fetal viral load could make possible to decrease symptomatology neonatal in a group of infected fetuses.

DETAILED DESCRIPTION:
The infection with cytomegalovirus (CMV) is the first cause of congenital neurological handicap of infectious origin. It is probable that the neonatal viral load is correlated with becoming of infected new-born babies. Among the active antiviral treatments against CMV, valacyclovir is the only whose fetal and maternal tolerance was evaluated during the pregnancy. Its harmlessness and its aptitude to decrease the CMV viral load justify to evaluate it in a study against placebo. Decrease the fetal viral load could make possible to decrease symptomatology neonatal in a group of infected fetuses.

To evaluate the effect of a treatment by valacyclovir injected per bone to the mother in the cases of proven fetal infection with CMV (positive PCR CMV in the amniotic liquid) and presenting cerebral extra echographic signs being able to be allotted to the infection.

The main objective is to observe in the treated group, a reduction in the number of unfavourable exits (symptomatic children at birth) and a reduction in the number of medical interruptions of pregnancy practised for fetal anomalies.

The secondary objective is a reduction in the treated group, of the CMV viral load in the blood of the cord taken at birth.

The attribution of the treatments will be carried out by drawing lot, according to a procedure in double blind as of the established diagnosis of the fetal infection. In the absence of reference treatment, a placebo will be employed in the reference group. The patients included will be thus placed in one of the 2 parallel groups. The observance will be evaluated. Taking into consideration our preliminary study, a difference of 20% between the 2 groups can be discounted. The number calculated of subjects to include in the test in order to guarantee a power of 80% to him is of 82 in each group. Recruitment will be carried out in a multicentric way. The necessary duration of inclusion will be 36 months

The comparison of the two treatments will be carried out on the composite principal criterion according to : proportion of pregnancies with unfavourable exit (symptomatic children at birth or medical interruptions of pregnancy practised for which has appeared cerebral echographic anomalies in connection with the fetal infection with CMV).

The secondary criteria of judgement will be : the viral load in the blood of the cord of the newborns infected in UTERO by CMV, the compliance and the criteria of tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years,
* Fetal Infection with CMV authenticated by the positivity of the research of the viral genome by PCR in the amniotic liquid,
* Echographic Assessment revealing at least one cerebral extra anomaly being able to be in connection with the infection with CMV,
* Absence of request for termination of pregnancy from the start,
* Acceptance of a strict follow-up by a Multi-field Center of Prenatal diagnosis and of an optimal observance of the founded treatment,
* Collection of the written assent to take part in the test.
* Affiliation with a mode of social security or equivalent

Exclusion Criteria:

* No affiliation with a mode of social security (profit or having right)
* Patient of less than 18 years,
* Patient presenting another pathology obstetrical or medical (in particular hepatic or renal) preexistent to tracking or contra-indicating the use of valacyclovir,
* Patients whose fetus does not present any echographic sign being able to be in connection with the infection with CMV,
* Patients whose fetus presents at least one cerebral echographic anomaly:IntraparenchymalVentriculomegaly measured with the ventricular crossroads ≥ 12mm

  * Hyperechogenicity periventricular
  * Hydrocephaly
  * Intra-ventricular adherence
  * Microcephaly
  * Increase cuts large retro-cerebellar cistern
  * Hypoplasia vermis
  * Intraparenchymal calcifications
  * Porencephaly
  * Lissencephaly
  * Cysts periventricular
  * Hypoplasia of the callous body
  * Signs of LENTICULO-striated vasculopathy
* Patient under any other active antiviral treatment against CMV,
* Patient taking part in another therapeutic test,
* Patient refusing to sign the enlightened assent,
* Patient formulating a request for medical interruption of pregnancy before inclusion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-09; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
pregnancies with unfavourable exit (symptomatic children at birth or medical interruptions of pregnancy practised for which has appeared cerebral echographic anomalies in connection with the fetal infection with CMV) at 24 hours | six months

SECONDARY OUTCOMES:
the viral load in the blood of the cord of the newborns infected in UTERO by CMV, the compliance at one month the criteria of tolerance | six months
the compliance at one month | six months
the criteria of tolerance | six months

CONTACTS AND LOCATIONS:
Overall Officials: Yves VILLE, PUPH, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hospital Necker Enfants Malades, Paris, France